CLINICAL TRIAL: NCT03143114
Title: Effect of Myomectomy for Intramural Myoma on Fertility Outcomes in Infertile Women: a Randomized Clinical Trial
Brief Title: Effect of Myomectomy for Intramural Myoma on Fertility Outcomes in Infertile Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WR3
Record Dates: First submitted 2017-05-04; First posted 2017-05-08 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Infertility; Fibroid
MeSH Terms: conditions — Infertility; Leiomyoma | interventions — Uterine Myomectomy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myomectomy (Experimental): Women will be subjected to laparotomy to remove the myomas
  Interventions: Procedure: Myomectomy
- Conservative management (No Intervention): Women will not be subjected to surgery (conservative management)

INTERVENTIONS:
Procedure: Myomectomy — Laparotomy then incision in the uterine wall to remove the myoma followed by closure of the uterine incision
  Arms: Myomectomy

SUMMARY:
The aim of this study is to evaluate the effect of myomectomy for intramural myomas on the fertility outcomes in infertile women.

DETAILED DESCRIPTION:
All women participating in the study will be randomly allocated into two groups; myomectomy group and conservative management group. Women in the myomectomy group will be subjected to laparotomy to remove the myomas while women in the conservative management group will not be subjected to surgery. Women in the myomectomy group will be asked to abstain from having sexual intercourse (or use a barrier contraception method) for 3 months after surgery then to start having regular fertility-oriented intercourse after that. Women in the conservative management group will be asked to immediately start having regular fertility-oriented intercourse. Women in both groups will be monitored form the time of starting regular intercourse and for one year for occurrence of clinical pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Infertility for at least one year.
* Presence of intramural myoma.
* Absence of any other cause of infertility as revealed by basic infertility work up including laparoscopy.

Exclusion Criteria:

* Age is < 20 or > 33 years.
* Symptomatic fibroid causing pelviabdominal swelling.
* Presence of > 2 myomas.
* Presence of a coexisting another type of myoma other than intramural myoma (e.g. submucosal, subserosal, cervical or ligamentary myoma).
* Presence of any other cause of infertility.

Ages: 20 Years to 33 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-05-15 (Actual); Primary Completion 2021-06-15 (Estimated); Study Completion 2021-06-15 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 6-8 weeks gestational age
  Number of clinical pregnancies (defined as presence of at least one intrauterine gestational sac with fetal pole and cardiac activity on TVS scan at 6-8 weeks gestational age) divided by the number of women

SECONDARY OUTCOMES:
Miscarriage rate | 12 weeks gestational age
  Number of first trimester miscarriages (before 12 weeks gestational age) divided by the number of clinical pregnancies

CONTACTS AND LOCATIONS:
Overall Officials: Waleed El-refaie, Dr, Principal Investigator — Port Said University; Khaled Samir, Dr, Study Director — Mansoura University; Mahmoud M Awad, Dr, Study Director — Mansoura University; Mohamed S Abdelhafez, Dr, Study Chair — Mansoura University
Locations (2):
- Egypt (2):
  - Obstetrics and Gynecology Department in Mansoura University Hospital, Al Mansurah, Dakahlia Governorate
  - Obstetrics and Gynecology Department in Mansoura University, Port Said

IPD SHARING:
Plan to Share IPD: Undecided